CLINICAL TRIAL: NCT00651118
Title: Randomized, Double-Blind Trial of MP29-02 Nasal Spray Compared to Placebo, Azelastine Hydrochloride Nasal Spray, and Fluticasone Propionate Nasal Spray in the Treatment of Patients With Seasonal Allergic Rhinitis
Brief Title: A Study to Evaluate the Safety and Effectiveness of a Nasal Spray to Treat Seasonal Allergies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP4002
Record Dates: First submitted 2008-03-28; First posted 2008-04-02 (Estimated); Results first posted 2012-09-26 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-08

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — azelastine; Fluticasone; MP29-02

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- fluticasone propionate (Active Comparator)
  Interventions: Drug: fluticasone propionate
- azelastineHcl/fluticasone propionate (Experimental)
  Interventions: Drug: azelastineHcl / fluticasone propionate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- azelastine Hcl (Active Comparator)
  Interventions: Drug: azelastine Hcl

INTERVENTIONS:
Drug: Placebo — placebo
  Arms: Placebo
Drug: azelastine Hcl — azelastine Hcl 548 mcg
  Other Names: azelastine
  Arms: azelastine Hcl
Drug: azelastineHcl / fluticasone propionate — azelastine Hcl 548 mcg / fluticasone propionate 200 mcg
  Other Names: MP29-02
  Arms: azelastineHcl/fluticasone propionate
Drug: fluticasone propionate — fluticasone propionate 200 mcg
  Other Names: fluticasone
  Arms: fluticasone propionate

SUMMARY:
The purpose of this study is to determine if two allergy medications (azelastine and fluticasone) are more effective than placebo or either medication alone (azelastine or fluticasone)

DETAILED DESCRIPTION:
This will be a Phase III, randomized, double-blind, placebo-controlled, parallel-group study in subjects with moderate-to-severe seasonal allergic rhinitis (SAR). The study will begin with a 7-day, single-blind, placebo lead-in period (Day -7 to Day 1). Subjects will be instructed to take placebo lead-in medication twice daily (1 spray per nostril), approximately every 12 hours. On Day 1, subjects who satisfy the symptom severity requirements and continue to meet all of the study inclusion/exclusion criteria will be randomized in a 1:1:1:1 ratio to receive 1 spray per nostril twice daily of MP29-02, azelastine hydrochloride, fluticasone propionate, or placebo nasal spray.

Efficacy will be assessed by the change from baseline in the subject-reported 12-hour reflective Total Nasal Symptom Score (TNSS). On Days 1 through 14, subjects will rate the instantaneous and reflective TNSS symptoms of sneezing, nasal congestion, runny nose, and nasal itching; the instantaneous and reflective total ocular symptom score (TOSS) symptoms of itchy eyes, watery eyes and eye redness; and the symptom of postnasal drip, twice daily (AM and PM) in a diary prior to the dose of study medication. Symptoms will be scored on a 0 to 3 scale (0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms, 3 = severe symptoms), such that the maximum daily symptom severity score will be 24 for the TNSS and 18 for the TOSS. Additional secondary efficacy variables will include reflective individual nasal and ocular symptom scores, as well as change from Baseline to Day 14 in the Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ).

Subjects ≥ 18 years of age will complete the RQLQ on Day 1 (prior to dosing) and Day 14. Subjects will return to the clinic on Day 7 for an interim evaluation. After completing the 2-week double-blind treatment period, subjects will return to the clinic on Day 14 (or at time of early termination) for an end-of-study evaluation. Safety and tolerability assessments will be made on Days 7 and 14. Tolerability will be evaluated by subject-reported adverse events (AEs), nasal examinations, and vital signs assessments.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 12 years of age and older with a 2 year history of moderate to severe seasonal allergic rhinitis
* Must be in generally good health
* Must meet minimum symptom requirements, as specified in the protocol
* Must be wiling and able to provide informed consent and to participate all study procedures
* Positive skin test to a prevalent spring allergen

Exclusion criteria:

* On nasal examination,the presence of nasal mucosal erosion, nasal ulceration or nasal septal perforation
* Nasal disease likely to affect the deposition of the medication or evaluation, such as sinus infection, nasal polyps or severe deviated septum
* Nasal or sinus surgery within the previous 6 months
* Chronic sinus infection (more than 3 per year)
* Planned travel outside the study area during the study period
* Use of any investigational drug within 30 days of the first visit
* Hypersensitivity (bad reaction) to azelastine hydrchloride nasal spray (Astelin), or fluticasone propionate nasal spray (Flonase)
* Women who are not using an acceptable method or birth control
* Women who are pregnant or nursing
* Upper respiratory tract infection such as common cold, flu, sinus infection within 2 weeks of first study visit
* Asthma or other lung diseases such as COPD. Mild asthma symptoms may be considered after consultation with the investigator
* Irregular heartbeat or other symptomatic heart conditions
* History of alcohol or drug abuse
* History of glaucoma
* Use of medications that could affect the study results

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 832 (Actual)
Dates: Start 2008-03; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lewis M. Fredane, MD, Study Director — Meda Pharmaceuticals
Locations (43):
- United States (43):
  - Allergy, Asthma and Immunology Associates, Scottsdale, Arizona
  - Clinical Research Center, Encinitas, California
  - Allergy Research Foundation, Los Angeles, California
  - Southern California Research, Mission Viejo, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Allergy and Asthma Medical Group and Research Center, San Diego, California
  - Bensch Research Associates, Stockton, California
  - Allergy and Asthma Clinical Research, Inc., Walnut Creek, California
  - Storms Clinical Research Institute, Colorado Springs, Colorado
  - Colorado Allergy and Asthma Centers, Denver, Colorado
  - Colorado Allergy and Asthma Centers, Lakewood, Colorado
  - Clinical Research Atlanta, Atlanta, Georgia
  - Aeroallergy Research Laboratories of Savannah, Savannah, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Sneeze, Wheeze and Itch Associates, Normal, Illinois
  - Kansas City Allergy and Asthma, Overland Park, Kansas
  - Northeast Medical Research Associates, North Dartmouth, Massachusetts
  - Clinical Research Institute, Minneapolis, Minnesota
  - Clinical Research Institute, Plymouth, Minnesota
  - The Clinical Research Center, St Louis, Missouri
  - Allergy, Asthma and Immunology Associates, Lincoln, Nebraska
  - The Asthma and Allergy Center, Papillion, Nebraska
  - Atlantic Research Center, Ocean City, New Jersey
  - Research Asthma, Sinus and Allergy Centers, Warren Township, New Jersey
  - AAIR Research Center, Rochester, New York
  - Island Medical Research, Rockville Centre, New York
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Bernstein Clinical Research Center, Cincinnati, Ohio
  - Allergy Clinic of Tulsa, Tulsa, Oklahoma
  - Allergy Asthma and Dermatology Research, Lake Oswego, Oregon
  - Allergy and Consultants of NJ/PA, Collegeville, Pennsylvania
  - Allergy and Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - Asthma and Allergy Research Associate, Upland, Pennsylvania
  - National Allergy, Asthma and Urticaria of Charleston, Charleston, South Carolina
  - East Tennesse Center for Clinical Research, Knoxville, Tennessee
  - Allergy and Asthma Associates, Austin, Texas
  - Allergy and Asthma Center of Austin, Austin, Texas
  - AARA Research Center, Dallas, Texas
  - Jane Lee, MD, PA Research Center, Dallas, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Sylvana Research Associates, San Antonio, Texas
  - Intermountain Clinical Research, Draper, Utah
  - Asthma, Inc., Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- MP29-02: MP29-02(fluticasone propionate 50 mcg / azelastine HCl 137 mcg) nasal spray
- Fluticasone Propionate: fluticasone propionate nasal spray
- Azelastine HCl: azelastine HCl nasal spray nasal spray
- Placebo: placebo nasal spray
Period: Overall Study
Arm/Group | MP29-02 | Fluticasone Propionate | Azelastine HCl | Placebo
Started | 207 | 207 | 208 | 210
Completed | 198 | 200 | 197 | 203
Not Completed | 9 | 7 | 11 | 7
Not completed — Adverse Event | 4 | 0 | 1 | 1
Not completed — Protocol Violation | 2 | 2 | 6 | 2
Not completed — Lost to Follow-up | 2 | 0 | 1 | 2
Not completed — administrative | 1 | 4 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MP29-02 | Fluticasone Propionate | Azelastine HCl | Placebo | Total
Number analyzed (Participants) | 207 | 207 | 208 | 210 | 832
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19 | 15 | 28 | 36 | 98
  Between 18 and 65 years | 183 | 185 | 172 | 166 | 706
  >=65 years | 5 | 7 | 8 | 8 | 28
Age Continuous [Mean (Standard Deviation); unit: years] | 37.3 (14.1) | 38.6 (14.1) | 36.2 (14.6) | 37.3 (16.0) | 37.3 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 127 | 130 | 133 | 532
  Male | 65 | 80 | 78 | 77 | 300
Region of Enrollment [Number; unit: participants]
  United States | 207 | 207 | 208 | 210 | 832

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 12-hour Reflective Total Nasal Symptom Score (rTNSS)
Description: change from baseline in 12-hour reflective(how did you feel in the last 12 hours) total nasal symptom score (rTNSS)consisting of nasal congestion,runny nose, itchy nose and sneezing scored twice daily (AM and PM) in diary cards for the entire 14 day study period.
  The measurement scale is 0 to 24.A reduction in symptom severity score is indicated by a negative value.The more negative value the better the result.
Time Frame: days 1 to 14
Population: intent to treat population (ITT)- must have had at least one post baseline efficacy assessment
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | MP29-02 | Fluticasone Propionate | Azelastine HCl | Placebo
Number analyzed (Participants) | 207 | 207 | 208 | 209
units on a scale | -5.6 (5.2) | -4.7 (4.7) | -4.2 (4.6) | -2.9 (3.9)

2. Secondary Outcome: Change From Baseline in 12 Hour Instantaneous Total Nasal Symptom Score (iTNSS)
Description: change from baseline in 12-hour instantaneous ( how do you feel now) total nasal symptom score (iTNSS)consisting of nasal congestion,runny nose, itchy nose and sneezing scored twice daily (AM and PM) in diary cards for the entire 14 day study period.
  The measurement scale is 0 to 24.A reduction in symptom severity score is indicated by a negative value.The more negative the value the better the result.
Time Frame: day 1 to day 14
Population: intent to treat population (ITT)- must have had at least one post baseline efficacy assessment
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Groups:
- MP29-02: fluticasone propionate 50 mcg / azelastine HCl 137 mcg nasal spray
- Azelastine HCl: azelastine HCl nasal spray
Arm/Group | MP29-02 | Fluticasone Propionate | Azelastine HCl | Placebo
Number analyzed (Participants) | 207 | 207 | 208 | 209
units on a scale | -5.2 (5.3) | -4.5 (4.7) | -4.0 (4.7) | -2.6 (4.1)

3. Secondary Outcome: Change From Baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ)at the End of 14 Days
Description: adult Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) scored at day 1(baseline) and at day 14.
  The scale is measured from a value of 0 to 24. A negative number corresponds to a change from baseline measurement.The more negative the value the better the result.
Time Frame: day 1 to day 14
Population: intent to treat( ITT)population (18 yrs of age or older) must have had at least one post baseline efficacy assessment
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | MP29-02 | Fluticasone Propionate | Azelastine HCl | Placebo
Number analyzed (Participants) | 176 | 184 | 174 | 169
units on a scale | -1.6 (1.4) | -1.6 (1.2) | -1.4 (1.1) | -0.9 (1.1)

ADVERSE EVENTS:
Arm/Group | MP29-02 | Fluticasone Propionate | Azelastine HCl | Placebo
Serious Adverse Events (participants affected / at risk) | 0/207 | 0/207 | 0/208 | 0/210
Other Adverse Events (participants affected / at risk) | 12/207 | 16/207 | 19/208 | 7/210
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MP29-02 (N=207) | Fluticasone Propionate (N=207) | Azelastine HCl (N=208) | Placebo (N=210)
dysgusia (Gastrointestinal disorders) | 5 (5) | 2 (2) | 7 (7) | 1 (1)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) | 4 (4) | 2 (2)
headache (Nervous system disorders) | 1 (1) | 5 (5) | 1 (1) | 3 (3)
nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 4 (4) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators participating in multicenter studies must agree not to present data gathered individually or by a subgroup of centers before the full, initial publication, unless this has been agreed to by all other investigators and Meda Pharmaceuticals.

Meda Pharmaceuticals requests that it receive copies of any intended communication reasonably in advance (at least 15 working days for an abstract or oral presentation and 45 working days for a manuscript)